CLINICAL TRIAL: NCT00339053
Title: The Effect of Immunonutrition on Outcome and Postoperative Recovery in Patients Undergoing Elective Surgical Repair of a Thoraco (Abdominal) Aneurysm Aorta
Brief Title: Immunonutrition and Thoracoabdominal Aorta Aneurysm Repair
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Antonius Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-04.01 TAA
Record Dates: First submitted 2006-06-19; First posted 2006-06-20 (Estimated); Last update posted 2006-10-23 (Estimated); Status verified 2006-10

CONDITIONS: Thoracic Aortic Aneurysm; Respiratory Insufficiency
Keywords: thoracic aortic aneurysm; immunonutrition; respiratory failure; lenght of stay ICU
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Respiratory Insufficiency | interventions — Immunonutrition Diet

INTERVENTIONS:
Drug: Immunonutrition ( Impact)

SUMMARY:
The purpose of this study is to determine whether immunonutrition and pre operative nutrition can reduce lenght of respirator support, lenght of stay in the ICU and incidence of post operative infections

DETAILED DESCRIPTION:
Elective surgical repair of a Thoraco (Abdominal) Aneurysm Aorta (T(A)AA) is associated with high mortality and morbidity. Important complications are renal failure, paraplegia and respiratory failure.

A retrospective study we performed also revealed high post operative infection rates and high incidence of respiratory failure.

Improving immune status may reduce the occurrence of infections due to immune chances. Immunonutrition may enhance the patient's immune system. Many clinical trials of immunonutrition in critically ill and surgical patients have been performed. In meta-analyses it has been shown that immunonutrition results in lower infections rates and shorter 'length of stay' in hospital after major surgery. Immunonutrition has not been studied yet in TAA(A) surgery. Controversy exists in septic patients.

We designed a prospective randomized placebo controlled trial to study the effect of immunonutrition on time on ventilatorsupport, lenght of stay in the intensive care unit and incidence of postoperative infections after TAA(A) surgery. Patients start with oral supplements besides their normal diet 5 days before surgery. After the operation, the nutrition is continued by protocol and administered by nasogastric tube until normal entral feeding is possible. The control group wil receive iso caloric and iso nitrogen nutrition.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective surgical repair Thoracic or thoraco abdominal aneurysm

Exclusion Criteria:

* endovascular repair
* pregnancy
* immunodeficiency
* use of immunosuppressiva
* chronic obstructive lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142
Dates: Start 2004-09; Study Completion 2008-01

PRIMARY OUTCOMES:
days on ventilator support
Lenght of stay ICU
Incidence infections

SECONDARY OUTCOMES:
biochemical markers organ failure
biochemical markers infectious parameters

CONTACTS AND LOCATIONS:
Overall Officials: Eric PA van Dongen, phD, Study Director — St. Antonius Hospital; Leon HJ Aarts, PhD, Study Chair — University Medical Center Groningen; leo Bras, MD, Study Director — St. Antonius Hospital; gert B Brunnekreef, MD, Principal Investigator — St. Antonius Hospital
Locations (1):
- st Antonius Hospital, Nieuwegein, Utrecht, Netherlands

REFERENCES:
- [Background] Coselli JS, LeMaire SA, Conklin LD, Koksoy C, Schmittling ZC. Morbidity and mortality after extent II thoracoabdominal aortic aneurysm repair. Ann Thorac Surg. 2002 Apr;73(4):1107-15; discussion 1115-6. doi: 10.1016/s0003-4975(02)03370-2. PMID 11996250
- [Background] Tepaske R, Velthuis H, Oudemans-van Straaten HM, Heisterkamp SH, van Deventer SJ, Ince C, Eysman L, Kesecioglu J. Effect of preoperative oral immune-enhancing nutritional supplement on patients at high risk of infection after cardiac surgery: a randomised placebo-controlled trial. Lancet. 2001 Sep 1;358(9283):696-701. doi: 10.1016/s0140-6736(01)05836-6. PMID 11551575
- [Background] Heyland DK, Novak F, Drover JW, Jain M, Su X, Suchner U. Should immunonutrition become routine in critically ill patients? A systematic review of the evidence. JAMA. 2001 Aug 22-29;286(8):944-53. doi: 10.1001/jama.286.8.944. PMID 11509059